CLINICAL TRIAL: NCT02220400
Title: Low Dose Ketamine Prevent the Postoperative Cognitive Dysfunction in Aged Patients Underwent Orthopaedic Surgery，a Randomized Control Double Blinded Multicenter Clinical Trail
Brief Title: Ketamine Prevent POCD
Acronym: KPPOCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KPPOCD
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Necrosis of Femoral Head; Knee Osteoarthritis
Keywords: Postoperative cognitive dysfunction; Ketamine; Surgery
MeSH Terms: conditions — Osteoarthritis, Knee; Postoperative Cognitive Complications | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Ketamine infusion group
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Normal saline infusion

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine

SUMMARY:
Previous study demonstrated that neuroinflammation induced by surgery is the main cause of the postoperative cognitive dysfunction. As an agonist of NMDA receptor, ketamine is proved to be an anti-inflammation agent. In present study investigators hypothesized that low dose ketamine would prevent the cognition decline after orthopedic surgery in aged patients.

ELIGIBILITY:
Inclusion Criteria:

* Elder than 60
* Easily communicated with Chinese
* Selected to kneel or hip replacement
* Agree to take part into this clinical trail

Exclusion Criteria:

* Existing cerebral disease， or have a history of neurological and psychiatric disease including AD, stroke and psychosis
* Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24
* Several audition or vision disorder
* Preoperative systolic Blood pressure over 190mmHg or diastolic pressure >100mmHg
* Existing a history of hyperthyroidism
* Patient with glaucoma
* Unwillingness to comply with the protocol or procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Short-term cognitive changes after surgery | The day before surgery and 7 days after surgery (or before leave hospital)
  Investigators would use mini-mental state examination(MMSE), Visual reproduction test,digit symbol，digit span,color trail test and Stroop color and word test for measuring the short-term cognitive changes of patients after surgery.
Long-term cognitive changes after surgery | The day before surgery and 2 months after surgery
  Investigators would use mini-mental state examination(MMSE), Visual reproduction test,digit symbol，digit span,color trail test and Stroop color and word test for measuring the long-term cognitive changes of patients after surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality